CLINICAL TRIAL: NCT02109666
Title: Long Term Experience With Abatacept in Routine Clinical Practice
Acronym: ACTION
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-151
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood (Spanish sub study only)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients treated with Abatacept: RA patients are treated with Abatacept IV according Summary of Product Characteristics (SmPC) in Europe and Product Monograph in Canada
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept
  Other Names: Orencia

SUMMARY:
The purpose of this study is to estimate the retention rate of Abatacept over 24 months in routine clinical practice in every participating country depending on the treatment line.

DETAILED DESCRIPTION:
Time Perspective: Other: Collection of the baseline data collected at Abatacept IV initiation, prospectively or retrospectively within maximum 3 months following the first administration. Other assessments are collected during the follow up period (maximum of 2 years by patient)

Biospecimen Retention: None Retained excepted for a local sub study (in Spain) where sample with DNA was retained

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or Female subjects of more than 18 years old
* Patients with a diagnosis of established moderate to severe active RA (as per the American College of Rheumatology revised criteria, 1987), who at their physician's discretion are treated with Abatacept according to the SmPC in Europe and the Product Monograph in Canada (initiating or already on treatment for maximum 3 months) and for whom baseline characteristics are available

Exclusion Criteria:

* Patients who are currently included in any interventional clinical trial in RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 2364 (Actual)
Dates: Start 2008-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Retention rate of Rheumatoid arthritis (RA) patients treated with Abatacept in routine clinical practice | Up to 24 months

SECONDARY OUTCOMES:
Major determinants of treatment discontinuation of RA patients treated with Abatacept | Up to 24 months
  Major determinants including prior RA treatment experience with biologics and clinical outcomes, such as Disease Activity Score 28 (DAS28), Health Assessment Questionnaire-Disability Index (HAQ-DI), Clinical Disease Activity Index (CDAI), Simplified Disease Activity Index (SDAI) and their derived criteria
Distribution of time-to-discontinuation of Abatacept therapy for each major determinant of treatment discontinuation, overall and depending on the treatment line | Up to 24 months
Association of prior RA treatment experience and clinical outcomes during the treatment course with patient reported outcomes (Patient satisfaction, Pain, Patient's Global Assessment) | Up to 24 months
Summary of treatment experience and outcomes after switching to a biologic or conventional Disease Modifying Anti-Rheumatic Drugs (DMARD) for patients who discontinue Abatacept therapy | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- Local Institution, Salzburg, Austria
- Local Institution, Ghent, Belgium
- Local Institution, St. John's, Newfoundland and Labrador, Canada
- Local Institution, Prague, Czechia
- Local Institution, Holbæk, Denmark
- Local Institution, Montpellier, France
- Local Institution, Heidelberg, Germany
- Local Institution, Crete, Greece
- Local Institution, Dublin, Dublin, Ireland
- Local Institution, Siena, Italy
- Local Institution, Amsterdam, Netherlands
- Local Institution, Seville, Spain
- Local Institution, Basel, Switzerland

REFERENCES:
- [Derived] Alten R, Behar C, Merckaert P, Afari E, Vannier-Moreau V, Ohayon A, Connolly SE, Najm A, Juge PA, Liu G, Rai A, Elbez Y, Lozenski K. Predicting abatacept retention using machine learning. Arthritis Res Ther. 2025 Feb 1;27(1):20. doi: 10.1186/s13075-025-03484-0. PMID 39893489
- [Derived] Alten R, Mariette X, Lorenz HM, Nusslein H, Galeazzi M, Navarro F, Chartier M, Heitzmann J, Poncet C, Rauch C, Le Bars M. Predictors of abatacept retention over 2 years in patients with rheumatoid arthritis: results from the real-world ACTION study. Clin Rheumatol. 2019 May;38(5):1413-1424. doi: 10.1007/s10067-019-04449-w. Epub 2019 Feb 21. PMID 30790095
- [Derived] Alten R, Mariette X, Lorenz HM, Galeazzi M, Cantagrel A, Nusslein HG, Chartier M, Elbez Y, Rauch C, Le Bars M. Real-world predictors of 12-month intravenous abatacept retention in patients with rheumatoid arthritis in the ACTION observational study. RMD Open. 2017 Dec 29;3(2):e000538. doi: 10.1136/rmdopen-2017-000538. eCollection 2017. PMID 29435360
- [Derived] Alten R, Burkhardt H, Feist E, Kruger K, Rech J, Rubbert-Roth A, Voll RE, Elbez Y, Rauch C. Abatacept used in combination with non-methotrexate disease-modifying antirheumatic drugs: a descriptive analysis of data from interventional trials and the real-world setting. Arthritis Res Ther. 2018 Jan 2;20(1):1. doi: 10.1186/s13075-017-1488-5. PMID 29329602
- [Derived] Alten R, Nusslein HG, Mariette X, Galeazzi M, Lorenz HM, Cantagrel A, Chartier M, Poncet C, Rauch C, Le Bars M. Baseline autoantibodies preferentially impact abatacept efficacy in patients with rheumatoid arthritis who are biologic naive: 6-month results from a real-world, international, prospective study. RMD Open. 2017 Feb 13;3(1):e000345. doi: 10.1136/rmdopen-2016-000345. eCollection 2017. PMID 28243468
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx